CLINICAL TRIAL: NCT02611687
Title: Double Blind, Multicentre, Randomized, Placebo-controlled Trial to Evaluate Safety and Efficacy of Pitolisant in Children From 6 to Less Than 18 Years With Narcolepsy With/Without Cataplexy, Followed by a Prolonged Open-label Period
Brief Title: Efficacy and Safety of Pitolisant in Pediatric Narcoleptic Patients With or Without Cataplexy, Double-blind Study Followed by a Prolonged Open-label Period
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bioprojet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P11-06/BF2.649; 2013-001506-29 (EudraCT Number)
Record Dates: First submitted 2015-11-16; First posted 2015-11-23 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Narcolepsy With Cataplexy; Narcolepsy Without Cataplexy
MeSH Terms: conditions — Narcolepsy | interventions — pitolisant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pitolisant (Experimental): tablet, oral, once a day.
  Interventions: Drug: pitolisant
- placebo (Placebo Comparator): tablet, oral, once a day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: pitolisant — Tablet
  Other Names: BF2.649
  Arms: pitolisant
Drug: Placebo — Tablet
  Arms: placebo

SUMMARY:
The purpose of this multicenter double blind study is to assess efficacy and safety of Pitolisant versus placebo in paediatric Narcoleptic patients with or without cataplexy.

ELIGIBILITY:
Inclusion Criteria:

* Male and female children from 6 to less than 18 years of age suffering from narcolepsy with or without cataplexy - ICSD-3 criteria (narcolepsy type 1 and 2).
* PDSS
* Patients should be free of non-authorized medication, in particular psychostimulant treatments as from the screening visit onwards.
* Parents - and patients old enough to understand who have expressed a willingness to participate in the study, who have signed and dated the informed consent form prior to beginning protocol required procedures.
* In the opinion of the investigator, the patient must have adequate support to comply with the entire study requirements as described in the protocol (e.g., transportation to and from trial site, self rating scales and diaries completion, drug compliance, scheduled visits, tests).

Exclusion Criteria:

* Any other conditions that can be considered the primary causes of EDS.
* Cataplectic patients treated by anticataplectics which are not under a stable treatment at the time of inclusion.
* Patients treated for cataplexy or any other pathology, by tricyclic antidepressants.
* Any significant abnormality of the electrocardiogram and particularly Fridericia's QTc interval.
* Patients with significant abnormality or clinical laboratory results.
* Psychiatric and neurological disorders in the investigator's opinion, would preclude the patient's participation and completion of this trial or comprise reliable representation of subjective symptoms.
* Active clinically significant illness, including unstable cardiovascular, endocrine, neoplastic, gastrointestinal, haematological, hepatic, immunologic, metabolic, neurological (other than narcolepsy/cataplexy), pulmonary, and/or renal disease which could interfere with the study conduct or counter-indicate the study treatments or place the patient at risk during the trial or compromise the study objectives.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 110 (Actual)
Dates: Start 2016-06-06 (Actual); Primary Completion 2021-04-03 (Actual); Study Completion 2025-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Plazzi, MD, Study Chair — Dipartimento di Scienze Biomediche e Neuromotorie Alma Mater Studiorum - Università di Bologna
Locations (11):
- Terveystalo Helsinki Uniklinikka, Helsinki, Finland
- France (3):
  - Hôpital Femme-Mère-Enfant, Bron
  - Hôpital Gui de Chauliac, Montpellier
  - Hôpital Robert Debré, Paris
- Università di Bologna, Bologna, Italy
- Polikliniek Heemstede Neurologist-Somnologist, Heemstede, Netherlands
- Russia (5):
  - Scientific-Research Medical Complex "Your Health", Kazan'
  - I.M. Sechenov First Moscow State Medical University, Moscow
  - V.M. Behterev National Medical Research Psychiatry and Neurology Center, Saint Petersburg
  - Samara Regional Clinical Hospital, Samara
  - N.I. Balaban Crimea Repiblic Clinical Psychiatric Hospital No. 1, Simferopol

REFERENCES:
- [Derived] Dauvilliers Y, Lecendreux M, Lammers GJ, Franco P, Poluektov M, Causse C, Lecomte I, Lecomte JM, Lehert P, Schwartz JC, Plazzi G. Safety and efficacy of pitolisant in children aged 6 years or older with narcolepsy with or without cataplexy: a double-blind, randomised, placebo-controlled trial. Lancet Neurol. 2023 Apr;22(4):303-311. doi: 10.1016/S1474-4422(23)00036-4. PMID 36931805

RESULTS

PARTICIPANT FLOW:
Period: Double-blind Period (0 to 8 Weeks)
Arm/Group | Pitolisant | Placebo
Started | 72 | 38
Completed | 70 | 37
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1
Period: Open-label Period (0 to >11 Months)
Arm/Group | Pitolisant | Placebo
Started | 70 (Participants having recieved pitolisant or placebo during the double-blind period of the study are treated with pitolisant in the open-label period) | 36 (All patients in open-label period are treated with pitolisant)
Completed | 39 (The open-label period is ongoing) | 21
Not Completed | 31 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pitolisant | Placebo | Total
Number analyzed (Participants) | 72 | 38 | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 72 | 38 | 110
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.0 (3.0) | 12.5 (3.0) | 12.9 (3.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 14 | 49
  Male | 37 | 24 | 61
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 72 | 38 | 110
Region of Enrollment [Number; unit: participants]
  Netherlands | 3 | 2 | 5
  Finland | 1 | 1 | 2
  Italy | 17 | 9 | 26
  France | 19 | 9 | 28
  Russia | 32 | 17 | 49

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate the Efficacy of Pitolisant in Reducing Residual Excessive Daytime Sleepiness (EDS), Ullanlinna Narcolepsy Scale Score.
Description: Changes in EDS measured by the Ullanlinna Narcolepsy Scale Score (UNS) from baseline (mean of two pre-treatment measures) to the end of double-blind period (mean of the last two measures).
  The UNS is an 11-item scale used to measure the intensity and frequency of symptoms of narcolepsy (EDS and cataplexy). The total score varies from 0 to 44, with higher scores denoting greater narcoleptic tendencies.
Time Frame: 8 weeks
Population: Full Analysis Set
Measure: Geometric Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pitolisant | Placebo
Number analyzed (Participants) | 72 | 38
score on a scale | -6.29 (1.14) | -2.60 (1.35)

2. Secondary Outcome: To Evaluate the Efficacy of Pitolisant in Reducing Residual Excessive Daytime Sleepiness (EDS), Pediatric Daytime Sleepiness Scale.
Description: Changes in EDS measured by the Pediatric Daytime Sleepiness Scale (PDSS) from baseline (mean of two pre-treatment measures) to the end of double-blind period (mean of the last two measures).
  The PDSS total score can range from 0 and 32 and a score >13 is considered abnormal sleepiness.
Time Frame: 8 weeks
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pitolisant | Placebo
Number analyzed (Participants) | 72 | 38
score on a scale | -5.53 (0.66) | -2.11 (0.89)

3. Secondary Outcome: To Evaluate the Efficacy of Pitolisant in Reducing Residual Excessive Daytime Sleepiness (EDS), Ullanlinna Narcolepsy Scale-Cataplexy Subscore .
Description: Changes in EDS measured by Ullanlinna Narcolepsy Scale-Cataplexy Subscore (UNS-CTP) in patients with type 1 narcolepsy from baseline (mean of two pre-treatment measures) to the end of double-blind period (mean of the last two measures).
  This subscore is defined as the sum of the first 4 items of the UNS, UNS-CTP subscore ranges from 0 to 16, with higher scores indicating more severe symptoms.
Time Frame: 8 weeks
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pitolisant | Placebo
Number analyzed (Participants) | 61 | 29
score on a scale | -2.88 (0.44) | -1.12 (0.64)

ADVERSE EVENTS:
Time Frame: 8 to 13 weeks (up to 4 weeks prior randomization, 8 weeks double-blind period and 1 week single-blind period)
Description: Other Adverse Events, reported with frequency threshold of 5%, are the most common Treatment Emergent Adverse Events.
  The open-label period of the study is ongoing, results of the open-label period will be available after completion of the study.
  Some patients did not receive the correct planned treatment, the safety analyses were performed by actual treatment group: 73 patients in the pitolisant group and 37 patients in the placebo group.
Arm/Group | Pitolisant | Placebo
All-Cause Mortality (participants affected / at risk) | 0/73 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/73 | 0/37
Other Adverse Events (participants affected / at risk) | 15/73 | 11/37
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pitolisant (N=73) | Placebo (N=37)
Headache (Nervous system disorders) | 14 (24) | 3 (4)
Insomnia (Psychiatric disorders) | 5 (5) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 3 (5)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-09-30): https://cdn.clinicaltrials.gov/large-docs/87/NCT02611687/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-15): https://cdn.clinicaltrials.gov/large-docs/87/NCT02611687/SAP_001.pdf